CLINICAL TRIAL: NCT06757829
Title: Pulmonary Functions in Sickle Cell Disease: Response of Adding Acu-TENS to Inspiratory Muscle Training
Brief Title: Pulmonary Functions in Sickle Cell Disease: Response to Acu-TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00014233-17
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): sickle cell disease patients whose number will be 20 patients will be trained with IMT (threshold inspiratory muscle training) and treated with AC-tens. The number of sessions per week will be three sessions for IMT or AC-tens for 12 weeks. the IMT will be performed for six sets of respiratory training cycles and the set will contain 10 respiratory cycles. Also the session of AC-tens will be 45 minute on bilateral Ex-B1 acupoint. the parameters of AC-tens will be four hertz and 200 microsecond pulse duration.
  Interventions: Behavioral: inspiratory muscle training and acupucnture like transcutanoeus electrical nerve stimulation
- Group II (Active Comparator): sickle cell disease patients whose number will be 20 patients who will trained with IMT (threshold inspiratory muscle training). The number of sessions per week will be three sessions for IMT for 12 weeks. the IMT will be performed for six sets of respiratory training cycles and the set will contain 10 respiratory cycles.
  Interventions: Behavioral: inspiratory muscle training

INTERVENTIONS:
Behavioral: inspiratory muscle training and acupucnture like transcutanoeus electrical nerve stimulation — sickle cell disease patients whose number will be 20 patients will be trained with IMT (threshold inspiratory muscle training) and treated with AC-tens. The number of sessions per week will be three sessions for IMT or AC-tens for 12 weeks. the IMT will be performed for six sets of respiratory training cycles and the set will contain 10 respiratory cycles. Also the session of AC-tens will be 45 minute on bilateral Ex-B1 acupoint. the parameters of AC-tens will be four hertz and 200 microsecond pulse duration.
  Arms: group I
Behavioral: inspiratory muscle training — sickle cell disease patients whose number will be 20 patients who will trained with IMT (threshold inspiratory muscle training). The number of sessions per week will be three sessions for IMT for 12 weeks. the IMT will be performed for six sets of respiratory training cycles and the set will contain 10 respiratory cycles.
  Arms: Group II

SUMMARY:
pulmonary complications are common in sickle cell disease patients. Respiratory training using inspiratory muscle trainer (IMT) is usually a good choice to improve these complications. Recently, acupuncture like transcutaneous electrical nerve stimulation (AC-tens) may also improve these complications.

DETAILED DESCRIPTION:
sickle cell disease patients whose number will be forty patients will be divided to group I who will trained with IMT (threshold inspiratory muscle training) and treated with AC-tens (the number of patients will be 20) or group II who will trained with IMT (the number of patients will be 20) . The number of sessions per week will be three sessions for IMT or AC-tens for 12 weeks. the IMT will be performed for six sets of respiratory training cycles and the set will contain 10 respiratory cycles. Also the session of AC-tens will be 45 minute on bilateral Ex-B1 acupoint. the parameters of AC-tens will be four hertz and 200 microsecond pulse duration.

ELIGIBILITY:
Inclusion Criteria:

* sickle cell disease patients
* non obese patients

Exclusion Criteria:

* patients with any systemic or chest or renal or hepatic or neurological diseases
* women with lactation or pregnancy
* patients atacks of vasoocclusive crisis

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
FEV1/FVC ratio | it will be assessed after12 weeks
  will be measured by spirometry

SECONDARY OUTCOMES:
forced expiratory volume at the first second of expiration | it will be assessed after12 weeks
  will be measured by spirometry
forced vital capacity | it will be assessed after12 weeks
  will be measured by spirometry
six minute walk distance | it will be assessed after12 weeks
  it will be a measure of physical capacity
physical summary of short form 36 | it will be assessed after12 weeks
  it is a questionnaire measure of quality of life
mental summary of short form 36 | it will be assessed after12 weeks
  it is a questionnaire measure of quality of life
right diaphragmatic excrusion | it will be measured after 12 weeks
  it will be assessed by ultrasonography
left diaphragmatic excrusion | it will be measured after 12 weeks
  it will be assessed by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt